CLINICAL TRIAL: NCT00099190
Title: A Phase Ib Safety and Pharmacokinetic Study of ARQ 501 in Combination With Docetaxol in Adult Patients With Locally Advanced or Metastatic Carcinoma
Brief Title: ARQ 501 in Combination With Docetaxel in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-111
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Carcinoma
Keywords: cancer; solid tumor; advanced solid tumor
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — beta-lapachone

INTERVENTIONS:
Drug: ARQ 501

SUMMARY:
The purpose of this study is to determine the safety of ARQ 501 in combination with docetaxel in patients with advanced or metastatic cancer. In addition, the study is designed to observe the potential the combination of ARQ 501 and docetaxel have in treating cancer.

DETAILED DESCRIPTION:
ARQ 501 has demonstrated activity in vitro against a wide range of solid tumors including lung, colorectal, breast, prostate, pancreatic, ovarian, and myeloma. To date, no histological cancer type studied appears inherently resistant to treatment with ARQ 501. In animal xenograft models of human tumors, ARQ 501 monotherapy has been effective in treating ovarian, colon, prostate, and breast cancer. When used in combination with taxane therapy, ARQ 501 has demonstrated efficacy in treating a variety of human cancers, including ovarian, breast, and colon.

This study is designed to explore whether the addition of ARQ 501 to a once every three week schedule of docetaxel is a safe and tolerable regimen. The study is designed to collect safety and pharmacokinetic data on the combination regimen and to measure the antitumor activity observed in patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed diagnosis of a locally advanced or metastatic carcinoma. (Patients may have either measurable or nonmeasurable disease.)
* Be ≥18 years old.
* Must not be eligible for therapy of higher curative potential.
* Have a Karnofsky Performance Status (KPS) of ≥70%.
* Have an estimated life expectancy of ≥12 weeks.
* Be male or non-pregnant, non-lactating female patients. Patients who are fertile agree to use an effective barrier method of birth control (e.g., latex condom, diaphragm, or cervical cap) to avoid pregnancy.
* Have a negative serum or urine pregnancy test within 7 days prior to the first dose of study drug (if patient is a female of childbearing potential).
* Sign a written informed consent document.
* Have adequate organ function as determined per protocol defined laboratory value

Exclusion Criteria:

* Have received previous treatment with ARQ 501.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Are pregnant or lactating.
* Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
* Have received any chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational, within 2 weeks of treatment in this study.
* Have not recovered from acute toxicity of all previous therapy prior to enrollment.
* Have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Have symptomatic or untreated central nervous system (CNS) metastases.
* Have a known severe hypersensitivity to docetaxel or drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of ARQ 501 in combination with docetaxel

SECONDARY OUTCOMES:
Collect information regarding antitumor activity of ARQ 501 in combination with docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: C. Casey Cunningham, MD, Principal Investigator — Mary Crowley Medical Research Center
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States